CLINICAL TRIAL: NCT03096574
Title: Respiratory Syncytial Virus (RSV) and Vaccination in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); St George's Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS project ID: 220968
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Respiratory Syncytial Virus (RSV); Maternal Vaccine Exposure; Attitude
Keywords: Respiratory Syncytial Virus (RSV); Maternal vaccination; Attitudes; Pregnancy
MeSH Terms: conditions — Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant women: * Over the age of 16
  * Under the care of staff working in: University Hospital Southampton NHS Foundation Trust, St Georges Healthcare NHS Trust, Oxford University Hospitals NHS Foundation Trust or University Hospitals Bristol NHS Foundation Trust
  * Able to read and write in English and give fully informed consent
  Interventions: Other: Questionnaire
- Maternity healthcare professionals: * Over the age of 18
  * Working in obstetrics or midwifery who regularly care for women in pregnancy at University Hospital Southampton NHS Foundation Trust, St Georges Healthcare NHS Trust, Oxford University Hospitals NHS Foundation Trust or University Hospitals Bristol NHS Foundation Trust
  * Able to read and write in English and give fully informed consent
- UK General Practitioners: * Fully-qualified general practitioners practicing in the UK
  * Able to read and write in English and give fully informed consent

INTERVENTIONS:
Other: Questionnaire — The participants will be approached by a member of the study team and, following recruitment, participants will be asked to fill in a short paper or online questionnaire. Our estimated time for completion is 5-10 minutes, and this time will be stated at the start of the questionnaire. Having completed the questionnaire they will be free to leave without further follow up, and given the contact details of the investigators/research governance office whom they can contact if they have further questions or concerns.
  Groups: Pregnant women

SUMMARY:
Respiratory Syncytial Virus (RSV) is the leading cause of chest infections (pneumonia and bronchiolitis) in young children, and is a major cause of admission to hospital and childhood death worldwide. One possible way to protect the mother and young infant from RSV infection is a vaccine given to women during pregnancy (maternal vaccination), which would pass protection to their unborn child. This may help to prevent RSV in the child's first few months of life when they are most vulnerable to infection.

There are two main aims to this study:

1. To pre-emptively gauge the knowledge of RSV and potential acceptability of such vaccines amongst pregnant women and healthcare staff working in midwifery and obstetrics, as well as their attitudes (facilitators and barriers) to being involved in hypothetical future research trials.
2. We also wish to gauge the attitudes to routinely recommended vaccines in pregnancy (pertussis and influenza)

The investigators propose to undertake a questionnaire-based study of randomly selected pregnant women and healthcare staff (over 16 years of age) at English teaching hospitals and GP practices. Pregnant women attending for ward reviews or antenatal clinics will approached and asked to complete an anonymous paper questionnaire lasting around 10 minutes. Healthcare staff will be approached in person, or via email, and asked to complete a slightly different questionnaire lasting around 5-10 minutes. No follow up will take place. Using statistical software, the investigators hope to identify factors that might affect patients' understanding of RSV and attitudes to being involved in hypothetical future trials and receiving routine vaccination

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is a very common virus that causes infection of the airways and lungs. It is the leading cause of chest infections (pneumonia and bronchiolitis) in young children, and is a major cause of admission to hospital and childhood death worldwide. Lots of research trials are being done into ways of preventing and treating RSV, however there is still no RSV vaccine approved for routine use. One possible way to protect the mother and young infant from RSV infection is a vaccine given to women during pregnancy, which would pass protection to their unborn child. This may help to prevent RSV in the child's first few months of life when they are most vulnerable to infection. There are two vaccines that are currently being tested in pregnant women around the world, including the UK.

There are two main aims to this study:

1. To pre-emptively gauge the knowledge of RSV and potential acceptability of such vaccines amongst pregnant women and healthcare staff working in midwifery and obstetrics, as well as their attitudes (facilitators and barriers) to being involved in hypothetical future research trials.
2. We also wish to gauge the attitudes to routinely recommended vaccines in pregnancy (pertussis and influenza)

The investigators propose to undertake a questionnaire-based study of randomly selected pregnant women and healthcare staff (over 16 years of age) at four English teaching hospitals. Pregnant women attending for ward reviews or antenatal clinics will approached and asked to complete an anonymous paper questionnaire lasting around 10 minutes. Healthcare staff will be approached in person, or via email, and asked to complete a slightly different questionnaire lasting around 5-10 minutes. No follow up will take place. Using statistical software, the investigators hope to identify factors that might affect patients' understanding of RSV and attitudes to being involved in hypothetical future trials and receiving routine vaccination

ELIGIBILITY:
1. Pregnant women

   Inclusion Criteria:
   * Over the age of 16
   * Under the care of staff working in: University Hospital Southampton NHS Foundation Trust, St Georges Healthcare NHS Trust, Oxford University Hospitals NHS Foundation Trust or University Hospitals Bristol NHS Foundation Trust
   * Able to read and write in English and give fully informed consent

   Exclusion Criteria:
   * Women in active labour
   * Women deemed acutely unwell or distressed
2. Maternity healthcare professionals

   Inclusion Criteria:
   * Over the age of 18
   * Working in obstetrics or midwifery who regularly care for women in pregnancy at University Hospital Southampton NHS Foundation Trust, St Georges Healthcare NHS Trust, Oxford University Hospitals NHS Foundation Trust or University Hospitals Bristol NHS Foundation Trust
   * Able to read and write in English and give fully informed consent
3. General practitioners

   * Fully-qualified and working in the UK
   * Able to read and write in English and give fully informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women and clinical staff at the four study sites
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Answers to questionnaires | Until data collection complete (December 2017)
  The answers to the questionnaires will be analysed using statistical software to assess their knowledge of RSV, and identify factors that might affect their understanding of RSV and attitudes to being involved in hypothetical future trials and receiving the RSV vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Jones, Study Chair — University Hospital Southampton NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Bristol University Hospitals, Bristol
  - St Georges Hospital, London
  - Oxford University Hospitals, Oxford
  - University Hosital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilcox CR, Calvert A, Metz J, Kilich E, MacLeod R, Beadon K, Heath PT, Khalil A, Finn A, Snape MD, Vandrevala T, Nadarzynski T, Coleman MA, Jones CE. Determinants of Influenza and Pertussis Vaccination Uptake in Pregnancy: A Multicenter Questionnaire Study of Pregnant Women and Healthcare Professionals. Pediatr Infect Dis J. 2019 Jun;38(6):625-630. doi: 10.1097/INF.0000000000002242. PMID 30418358
- [Derived] Wilcox CR, Bottrell K, Paterson P, Schulz WS, Vandrevala T, Larson HJ, Jones CE. Influenza and pertussis vaccination in pregnancy: Portrayal in online media articles and perceptions of pregnant women and healthcare professionals. Vaccine. 2018 Nov 29;36(50):7625-7631. doi: 10.1016/j.vaccine.2018.10.092. Epub 2018 Nov 3. PMID 30401620